CLINICAL TRIAL: NCT02336139
Title: A Phase II, Open-label, Single Arm, Multicentre, International Trial of Sofosbuvir (SOF) and GS-5816 for People With Chronic Hepatitis C Virus Infection and Recent Injection Drug Use
Brief Title: A Phase II Trial of Sofosbuvir (SOF) and GS-5816 for People With Chronic Hepatitis C Virus Infection and Recent Injection Drug Use
Acronym: SIMPLIFY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1309
Record Dates: First submitted 2015-01-04; First posted 2015-01-12 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sofosbuvir (SOF)/GS-5816 (Experimental): 12 weeks of Sofosbuvir (SOF)/GS-5816 (400mg/100mg) in an oral once-daily fixed dose combination
  Interventions: Drug: Sofosbuvir (SOF)/GS-5816

INTERVENTIONS:
Drug: Sofosbuvir (SOF)/GS-5816 — 12 weeks of Sofosbuvir (SOF)/GS-5816 (400mg/100mg) in an oral once-daily fixed dose
  Other Names: SOF/GS-5816

SUMMARY:
To evaluate the proportion of patients with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) following sofosbuvir/GS-5816 therapy for 12 weeks in people with chronic HCV infection and recent injection drug use.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have voluntarily signed the informed consent form.
2. 18 years of age or older.
3. Chronic HCV infection as defined by anti-HCV antibody or HCV RNA detection for greater than 6 months.
4. HCV RNA plasma ≥ 1000 IU/ml at Screening.
5. HCV genotypes 1-6.
6. Recent injecting drug use (previous 6 months).
7. Compensated liver disease.
8. Participants with Fibroscan >12 KPa or AFP >50 ng/mL must have an abdominal ultrasound or CT scan without evidence of hepatocellular carcinoma within 2 months prior to screening.
9. Negative pregnancy test at baseline (females of childbearing potential only).
10. All fertile males and females must be using effective contraception during treatment and during the 30 days after treatment end.

Exclusion Criteria:

1. History of any of the following:

   1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the participant treatment, assessment or compliance with the protocol; participants currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded.
   2. Clinical hepatic decompensation (i.e. ascites, encephalopathy or variceal haemorrhage)
   3. Solid organ transplant
   4. Malignancy within 5 years prior to screening, with exception of specific cancers that may have been cured by surgical resection (basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are also excluded.
   5. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
2. Screening ECG with clinically significant abnormalities
3. Any of the following lab parameters at screening:

   1. ALT > 10 x ULN
   2. AST > 10 x ULN
   3. Direct bilirubin > 1.5 x ULN
   4. Platelets < 50,0000/μL
   5. HbA1c > 8.5%
   6. Creatinine clearance (CLcr) < 60 mL/min
   7. Haemoglobin < 11 g/dL for females ; < 12 g/dL for males
   8. Albumin < 30g/L
   9. INR > 1.5 ULN unless subject has known haemophilia or is stable on an anticoagulant regimen affecting INR
4. Pregnant or nursing female.
5. HIV infection or HBV infection (HBcAb and HBsAg positive)
6. Use of prohibited concomitant medications as described in section 5.2
7. Chronic use of systemically administered immunosuppressive agents (e.g. prednisone equivalent > 10 mg/day)
8. Known hypersensitivity to GS-5816, sofosbuvir (SOF) or formulation excipients.
9. Therapy with any anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤6 months prior to the first dose of study drug.
10. Any investigational drug ≤6 weeks prior to the first dose of study drug.
11. Previous therapy with sofosbuvir (SOF) or an NS5A inhibitor prior to the first dose of study drug.
12. Ongoing severe psychiatric disease as judged by the treating physician.
13. Frequent injecting drug use that is judged by the treating physician to compromise treatment safety.
14. Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Sustained Virological Response (SVR12) | Week 24
  To evaluate the proportion of patients with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) following sofosbuvir (SOF)/GS-5816 therapy for 12 weeks in people with chronic HCV infection and recent injection drug use.

SECONDARY OUTCOMES:
Treatment adherence | Baseline to Week 12
  To evaluate the proportion of patients adherent to therapy (both on-treatment adherence and treatment discontinuation)
Impact of adherence on therapy (association between adherence and response to treatment ) | early (0-3 weeks), mid (4-7 weeks) and late (8-11 weeks) during therapy
  To evaluate the association between adherence and response to treatment [including an evaluation of the impact of early (0-3 weeks), mid (4-7 weeks) and late (8-11 weeks) missed doses on response to therapy]; Adehernce will be measure via a self report quesitonanire and pill counts via return of the weeekly blister packs. The impact of the number and timing of missed pills will be evaluated.
Factors associated with on-treatment adherence | Baseline to Week 12
  To evaluate factors associated with on-treatment adherence >90% and treatment discontinuation. Demographic and behavioural factors will be examined.
End of Treatment Response (ETR) (proportion of participants with undetectable HCV RNA at the end of treatment (ETR) | Week 12
  To evaluate the proportion of participants with undetectable HCV RNA at the end of treatment (ETR)
Safety and tolerability (number and type of adverse events and serious adverse events) | Baseline to Week 24
  To evaluate the number and type of adverse events and serious adverse events on treament and for 12 weeks post end of treatment
Change in drug use | Baseline to Week 12
  To evaluate the change in drug use during treatment
Change in mental health | Basleine to Week 12
  To evaluate the change in mental health during treatment
Change in health related quality of life | Baseline to Week 12
  To evaluate the change in health-related quality of life during treatment
Impact of mixed infection on treatment response | Baseline to Week 24
  To evaluate the rate of mixed HCV infection at baseline and among those with treatment non-response
Reinfection Rate | Week 108
  To evaluate the rate of HCV reinfection during and up to two years following treatment
Immunovirological factors associated with treatment clearance | Week 24
  To evaluate immunovirological factors associated with treatment clearance. We will evaluate cytokines and chemokines (e.g. interferon inducible protein 10), T-cell responses, viral evolution and genetic markers (e.g. inteferon lambda 4) that are potentially associated with treatment induced clearance
Utility of Dried Blood Spot (DBS) (method for monitoring HCV including treatment response) | Week 108
  To evaluate the utility of dried blood spot (DBS) as a simple method for monitoring HCV including treatment response. HCV RNA will be measured from DBS samples and then compared to HCV RNA levels measured using standard methods (EDTA Plasma samples and Roche Taqman)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Dore, MBBS PhD, Principal Investigator — Kirby Institute
Locations (1):
- The Kirby Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Cunningham EB, Hajarizadeh B, Amin J, Hellard M, Bruneau J, Feld JJ, Cooper C, Powis J, Litwin AH, Marks P, Dalgard O, Conway B, Moriggia A, Stedman C, Read P, Bruggmann P, Lacombe K, Dunlop A, Applegate TL, Matthews GV, Fraser C, Dore GJ, Grebely J. Reinfection Following Successful Direct-acting Antiviral Therapy for Hepatitis C Virus Infection Among People Who Inject Drugs. Clin Infect Dis. 2021 Apr 26;72(8):1392-1400. doi: 10.1093/cid/ciaa253. PMID 32166305
- [Derived] Artenie AA, Cunningham EB, Dore GJ, Conway B, Dalgard O, Powis J, Bruggmann P, Hellard M, Cooper C, Read P, Feld JJ, Hajarizadeh B, Amin J, Lacombe K, Stedman C, Litwin AH, Marks P, Matthews GV, Quiene S, Erratt A, Bruneau J, Grebely J. Patterns of Drug and Alcohol Use and Injection Equipment Sharing Among People With Recent Injecting Drug Use or Receiving Opioid Agonist Treatment During and Following Hepatitis C Virus Treatment With Direct-acting Antiviral Therapies: An International Study. Clin Infect Dis. 2020 May 23;70(11):2369-2376. doi: 10.1093/cid/ciz633. PMID 31300820
- [Derived] Grebely J, Dalgard O, Conway B, Cunningham EB, Bruggmann P, Hajarizadeh B, Amin J, Bruneau J, Hellard M, Litwin AH, Marks P, Quiene S, Siriragavan S, Applegate TL, Swan T, Byrne J, Lacalamita M, Dunlop A, Matthews GV, Powis J, Shaw D, Thurnheer MC, Weltman M, Kronborg I, Cooper C, Feld JJ, Fraser C, Dillon JF, Read P, Gane E, Dore GJ; SIMPLIFY Study Group. Sofosbuvir and velpatasvir for hepatitis C virus infection in people with recent injection drug use (SIMPLIFY): an open-label, single-arm, phase 4, multicentre trial. Lancet Gastroenterol Hepatol. 2018 Mar;3(3):153-161. doi: 10.1016/S2468-1253(17)30404-1. Epub 2018 Jan 6. PMID 29310928